CLINICAL TRIAL: NCT02096965
Title: Use of Tolvaptan to Reduce Urinary Supersaturation: a Pilot Proof of Principle Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, John Lieske, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 11-001780
Record Dates: First submitted 2014-03-24; First posted 2014-03-26 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Nephrolithiasis, Calcium Oxalate; Nephrolithiasis, Calcium Phosphate
Keywords: Calcium oxalate; Calcium phosphate; Kidney stone
MeSH Terms: conditions — Nephrolithiasis, Calcium Oxalate; Nephrolithiasis; Kidney Calculi | interventions — Tolvaptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tolvaptan first, then Placebo (Experimental): Tolvaptan twice daily in first intervention period and placebo twice daily in second intervention period. (after washout period)
  Interventions: Drug: Tolvaptan; Drug: Placebo
- Placebo first, then Tolvaptan (Experimental): Placebo twice daily in first intervention period and Tolvaptan twice daily in second intervention period. (after washout period)
  Interventions: Drug: Tolvaptan; Drug: Placebo

INTERVENTIONS:
Drug: Tolvaptan — Patients will receive daily dose of 45 mg (30 mg at 8 AM and 15 mg at 4 PM).
  Other Names: Samsca
Drug: Placebo — Patients will receive daily dose at 8 AM and at 4 PM.

SUMMARY:
In this study the investigators propose to use a daily dose of 45 mg (30 mg at 8 AM and 15 mg at 4 PM). This relatively small well-tolerated dose is likely to persistently increase urine volume and reduce urine supersaturation and to be well tolerated by patients with kidney stone disease and normal renal function (see below). The twice-daily (8 AM and 4 PM) regimen is designed to produce a maximal AVP inhibition on waking with a gradual fall-off of effect during the night. To this end, a higher dose is used in the morning, with a lower dose in the afternoon.

ELIGIBILITY:
Inclusion Criteria:

* History of calcium oxalate or calcium phosphate stone.
* Good renal function

Exclusion Criteria:

* History of hypo-or hypernatremia.
* History of hypotension or orthostatic dizziness.
* Clinical history of congestive heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in urinary calcium oxalate supersaturation (SS) | Baseline to 3 weeks
  Calcium oxalate (CaOx) SS is primary endpoint for CaOx stone formers.
Change in Calcium phosphate SS | Baseline to three weeks
  Calcium phosphate (CaPhos) SS is the primary endpoint for CaPhos stone formers.

CONTACTS AND LOCATIONS:
Overall Officials: John Lieske, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States